CLINICAL TRIAL: NCT07144358
Title: Effectiveness of Breastfeeding Arm Sling and Biological Feeding Position in Primiparous Women: A Randomized Controlled Trial
Brief Title: Effectiveness of Breastfeeding Arm Sling and Biological Feeding Position in Primiparous Womenl
Acronym: EBASBFP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Gul OZTAS (Other)
Responsible Party: Sponsor-Investigator, Hatice Gul OZTAS, DR., Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIU11
Record Dates: First submitted 2025-08-17; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Primiparous Women
Keywords: Breastfeeding; biological nurturing,; breastfeeding arm sling; midwifery
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Breastfeeding Arm Support group
  Interventions: Behavioral: Biological Feeding Position
- control group (Placebo Comparator): education
  Interventions: Behavioral: Biological Feeding Position

INTERVENTIONS:
Behavioral: Biological Feeding Position — Biological Feeding Position

SUMMARY:
Abstract

The World Health Organization (WHO) recommends that babies be fed exclusively with breast milk for the first six months after birth (World Health Organization, 2020). However, for women who are breastfeeding for the first time (primiparas), the breastfeeding process often presents both physical and psychological challenges. In recent years, technological and ergonomic solutions have been developed to support the breastfeeding process, and a new tool called a 'breastfeeding arm sling' is planned to be developed. This arm sling aims to support the mother's arm, allowing the baby to be positioned more stably and thus making the breastfeeding process more comfortable . On the other hand, the biological feeding position (laid-back breastfeeding) is an effective method that uses the effects of gravity to activate the baby's natural reflexes and allows the mother to breastfeed in a comfortable position . This study is a randomised controlled experimental study aimed at comparing the effects of the newly developed Breastfeeding Arm Support and the biological feeding position on breastfeeding in primiparous women. The research will be conducted with primiparous women who gave birth between September and December 2025 at the Women's Delivery Services 1 and 2 of Gaziantep Abdulkadir Yüksel State Hospital. Data will be collected through face-to-face interviews and questionnaire forms in the form of pre-tests and post-tests. The study includes two groups:

1. Group receiving the Breastfeeding Arm Support group (n = 44)
2. Group receiving the Biological Feeding Position (n = 44) Post-intervention post-tests will be administered to both groups, and the results will be compared.

DETAILED DESCRIPTION:
Breastfeeding is a fundamental life process for newborns in terms of nutrition, immunity and emotional bonding. The World Health Organization (WHO) recommends that babies be fed exclusively with breast milk for the first six months after birth . However, the breastfeeding process for primiparas is often accompanied by physical and psychological difficulties. Inability to achieve the correct breastfeeding position can lead to nipple cracks, inadequate nutrition for the baby, and decreased motivation to breastfeed .

In recent years, technological innovations and ergonomic support tools have been developed to improve the breastfeeding process. One of the ergonomic support tools used to facilitate the breastfeeding process is the breastfeeding arm sling. The breastfeeding arm sling aims to make the breastfeeding process more comfortable by supporting the mother's arm and ensuring that the baby is positioned more stably . In this regard, it is important to test new generation supportive breastfeeding equipment through evidence-based research.

On the other hand, the biological feeding position (laid-back breastfeeding) is a method that uses the effect of gravity to activate the baby's natural reflexes and allows the mother to breastfeed in a comfortable position. This position has been found to increase breastfeeding success, reduce nipple trauma, and facilitate milk flow, especially in primiparous women . However, there are limited studies in the literature suggesting that both methods can increase breastfeeding success.

This study aims to compare the effects of the breastfeeding support armrest and the biological feeding position on the breastfeeding process in primiparous women. Conducted within a randomised controlled design, this research aims to evaluate their effects on breastfeeding self-efficacy, breastfeeding success, and attitudes towards breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand Turkish well
* Applied within the first 72 hours after hospitalization
* Delivered a healthy newborn
* Age 18 years or older

Exclusion Criteria:

* Communication difficulties
* Inability to speak or understand Turkish

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 88 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Iowa Infant Feeding Attitudes Scale, | 48 hours
  developed by De La Mora and Russell (1999), was designed to assess women's attitudes toward breastfeeding and predict breastfeeding duration and infant feeding method selection. The scale consists of 17 items on a 5-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). Nine items in the scale contain negative statements about breastfeeding, while eight items contain positive statements about formula feeding. The scale's validity and reliability in Turkish were conducted by Ekşioğlu et al. (2016), and Cronbach's alpha was found to be 0.71 (Ekşioğlu et al., 2016).
Postnatal Breastfeeding Self-Efficacy Scale-Short Form Breastfeeding: | 2 day
  A 14-item short form of the 33-item scale, originally developed by Dennis and Faux9 to assess mothers' breastfeeding self-efficacy levels, was developed in 2003, and its Cronbach's alpha was found to be 0.94. Tokat Aluş and Okumuş18,19 found Cronbach's alpha to be 0.86 in the Turkish reliability and validity study of the short form of the Breastfeeding Self-Efficacy Scale, indicating its suitability for Turkish culture. In this study, the Cronbach's alpha value for the scale was 0.89. The Breastfeeding Self-Efficacy Short Form is a 5-point Likert-type scale (1 = Not at all confident to 5 = Always confident). The minimum score is 14, and the maximum score is 70. Higher scores indicate higher breastfeeding self-efficacy. The average administration time for the scale is 5-7 minutes.
LATCH | 2 day
  Breastfeeding Diagnostic Measurement Tool The LATCH Breastfeeding Diagnostic and Assessment Scale was developed by Jensen and colleagues in 1994 (Jensen, Wallace, and Kelsay 1994). The Turkish validity and reliability of the scale was conducted by Yenal and Okumuş in 2003 (Yenal and Okumuş 2003). The LATCH scale assesses the baby's attachment to the breast (L), audibility of swallowing (A), nipple type (T), nipple comfort (C), and the way the baby is held (H) (Jensen et al. 1994). Each item ranges from 0 to 2 points, with the lowest possible score being 0 and the highest being 10. The scale has no cut-off point. A high score indicates high breastfeeding success, while a low score indicates a need for breastfeeding support. In the most recent Turkish validity and reliability study of the scale, the Cronbach's alpha was reported as 0.95 (Yenal and Okumuş 2003).

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data because of institutional policies and protection of participant confidentiality.

REFERENCES:
- See also: Related Info — https://jer-nursing.org/jvi.aspx?pdir=jern&plng=eng&un=JERN-94547&look4=